CLINICAL TRIAL: NCT06465771
Title: Feasibility of a Youth-led NCD Risk Reduction Initiative in Selected Schools of Slums in Karachi, Pakistan: a Mixed-methods, pre-and Post-intervention Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Royal Society of Tropical Medicine and Hygiene (Other)
Responsible Party: Principal Investigator, Sabahat Naz, Senior Instructor, Aga Khan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 9763
Record Dates: First submitted 2024-05-27; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus; Cardiovascular Diseases; Cancer; Lung Diseases
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Neoplasms; Lung Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Youth-led NCD risk reduction initiative (Experimental): Students of grades 5 and 6 will receive NCD risk reduction intervention from youth (students of grades 9 and 10). The shared risk factors will include unhealthy diet, physical activity, and tobacco use. The NCDs will cover diabetes, cardiovascular disease, hypertension, and cancers.
  Interventions: Behavioral: Youth-led NCD risk reduction intervention

INTERVENTIONS:
Behavioral: Youth-led NCD risk reduction intervention — With the help of Youth (students of grades 9 and 10), their parents and other stakeholders, including teachers, headteachers, and canteen staff through qualitative interviews, we will develop an intervention focuses on NCD risk reduction among younger peers (students of grades 5 and 6). A nutritionist will train the youth on how to deliver the intervention among their younger peers.

SUMMARY:
The study will occur in ten selected schools within Azam Basti and Mehmoodabad, organized into five sequential phases. Phase I involves identifying NCD modifiable risk factors among younger peers (Classes 5 and 6 students) using structured diaries. Phase II includes qualitative interviews with youth (Classes 9 and 10 students), parents, and stakeholders to discuss intervention material and delivery. Phase III comprises a one-day workshop to co-create an intervention. Phase IV involves three-day training for youth to understand and deliver the intervention to their peers. Finally, Phase V assesses the intervention's feasibility using a pre-and post-test design approach.

ELIGIBILITY:
Inclusion Criteria:

1. Both government and private schools
2. Schools that have classes 1 to 10 in one boundary
3. Schools who agree to take part in the qualitative interviews
4. Schools that permit to engage youth, their parents, and younger peers in the study for ten months
5. For youth: Students of classes 9 and 10 (aged 14 to 16 years)
6. For younger peers: Students of classes 5 and 6 (9 to 12 years)
7. Students who provide written informed assent followed by parental consent
8. Parents of youth and other stakeholders, including head teachers, schoolteachers, and canteen staff who provide written informed consent

Exclusion Criteria:

1. Schools currently enrolled in any NCD-related intervention program or any similar program during the last six months
2. For youth: Having any severe or chronic medical condition or disability that restricts active participation of students in the intervention co-creation and delivery

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The compliance of delivering the intervention in schools using a fidelity checklist | Three months
  Once the intervention will be finalized, a fidelity checklist will be developed and used to assess adherence to the intervention delivery. It will be reported as if the intervention is delivered completely, partially, or incomplete based on each component of the intervention
The recruitment and attrition rates for schools and children | Ten months
  The recruitment and attrition rates will be assessed by reporting the frequencies and percentages of schools and children (youth and younger peer) enrolled and retained in the study.
The rate for completing the structured diaries for diet, physical activity, and tobacco use at pre-and post-intervention assessments | Ten months
  The frequencies and percentages of children completing the structured diaries for diet, physical activity, and tobacco use at pre-and post-intervention assessments will be reported.
The change in the frequency and percentages of risk factors, including unhealthy diet, physical inactivity, and tobacco use at post-intervention compared to the baseline using a structured diary | Ten months
  The change in the frequency and percentages of risk factors, including unhealthy diet, physical inactivity, and tobacco use at post-intervention compared to the baseline will be reported. The information will be collected through structured diaries at baseline and after the intervention is delivered. The students will complete the diary for four days before and after the intervention.

REFERENCES:
- [Derived] Naz S, Ilyas M, Iqbal R. Feasibility of co-creating and delivering a youth-led noncommunicable diseases risk reduction intervention in schools of slums in Karachi, Pakistan: protocol for a mixed-methods, pre- and post-intervention study. Pilot Feasibility Stud. 2025 Jun 2;11(1):76. doi: 10.1186/s40814-025-01662-0. PMID 40457417